CLINICAL TRIAL: NCT00221897
Title: Diagnostic Innovations in Glaucoma Study
Acronym: DIGS
Status: Recruiting | Type: Observational
Sponsor: University of California, San Diego (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Principal Investigator, Linda Zangwill, Principal Investigator, University of California, San Diego
Other Study IDs: EY08208; EY11008, EY027510; R01EY027510 (NIH)
Record Dates: First submitted 2005-09-14; First posted 2005-09-22 (Estimated); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Primary Open Angle Glaucoma; Myopia
Keywords: Primary open angle glaucoma; Glaucoma/pathology; Glaucoma/physiopathology; Nerve Fibers/pathology; Risk factors glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle; Myopia; Glaucoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Healthy individuals: healthy controls with or without myopia
- Persons at risk for or with primary open angle glaucoma: with or without myopia with a diagnosis of glaucoma, glaucoma suspect and ocular hypertension

SUMMARY:
The overarching goal of our research study is to evaluate changes in visual function and optic nerve topography (the structure of the back of the eye) in patients with glaucoma (increased susceptibility to pressure inside the eye that can cause loss of vision) or those with an increased risk of developing the disease. The purpose of this study is to determine the best methods for detecting the presence or progression (worsening over time) of glaucoma in patients with and without myopia and its effects on daily and visual function and quality of life. With several sources of NIH and foundation funding over the last twenty years we have designed a robust research protocol to address the most challenging aspects of glaucoma management. The most recent focus of this research is 1) to improve our ability to detect open angle glaucoma in individuals with myopia and in individuals of European and African descent, 2) to determine whether monitoring of the retinal vasculature with new optical imaging instruments can improve glaucoma management and elucidate the pathophysiology of the disease, and 3) to differentiate between age-related changes and glaucomatous progression.

The grants supporting this project include 3 NIH funded studies, 1) the University of California, San Diego UCSD -based "Diagnostic Innovations in Glaucoma Study" (DIGS funded since 1995): 2) the "African Descent and Glaucoma Evaluation Study" (ADAGES funded since 2002), 3) the Brightfocus Foundation National Glaucoma Research Program and 4) the UCSD-based "Diagnosis and Monitoring of Glaucoma with Optical Coherence Tomography Angiography" (funded since 2018). The ADAGES is a multi-center study with data collection also conducted at 2 other academic sites, the University of Alabama at Birmingham, and Columbia University.

Enrolled healthy participants, glaucoma suspects and glaucoma patients are generally asked to return for two or more visits a year for several years. We then analyze whether the glaucoma patients are progressing and what factors influence their glaucoma status compared to healthy subjects and individuals suspected of having glaucoma.

DETAILED DESCRIPTION:
The Diagnostic Innovation in Glaucoma Study (DIGS) and ADAGES are longitudinal studies in which participants with or without myopia are examined approximately biannually, in most cases. Healthy controls with or without myopia are examined once, in most cases. The ADAGES recruitment and testing of individuals of African descent is an independently funded multi-center (including UCSD, Columbia University, and University of Alabama, Birmingham) study, which follows the same study protocol as the DIGS to ensure that the data from both studies can be analyzed together. This harmonization of protocols leverages the advantages of both DIGS by increasing the sample sizes to address the unique hypotheses of each study.

All participants must be 18 years old or older. Participants with or without myopia will be required to have at least one eye with open angles, best corrected visual acuity of 20/40 or better to be included. Participants taking a medication known to affect visual field sensitivity and eyes with a history of intraocular surgery (except uncomplicated glaucoma and cataract surgery), a secondary cause of elevated intraocular pressure, a coexisting intraocular disease affecting visual field, or a problem other than glaucoma affecting color vision may be excluded.

Most of the extensive testing completed for these visits can be considered standard of care, but for clinical care all tests are not generally all done at the same patient visit with the variety of instruments included in this research project. The following tests can be considered standard of care: medical history, blood pressure and heart rate, height and weight, visual acuity testing near acuity testing, low contrast sensitivity testing, slit lamp biomicroscopy (including gonioscopy), measurements of intraocular pressure with contact and non-contact tonometry, corneal thickness measurement (pachymetry), corneal elasticity measured using non-contact tonometry, interocular axial length, corneal curvature, anterior chamber depth measurements (all measured using intraocular lens IOL master), dilated fundoscopy, stereoscopic ophthalmoscopy of the optic disc with a 78 D lens, color vision testing, standard automated perimetry, optical coherence tomography (OCT) and photography.

There is currently no end date to the study, as the follow-up will continue as long as the research is supported.

The time involved is usually 2-4 visits per year of approximately 2-5 hours each.

DIGS Positional Study Subjects will also be given the opportunity to participate in the following additional auxiliary study. The DIGS Positional Study will allow subjects to participate in an ancillary study. Participation in this ancillary study includes imaging of the eyes using Optical Coherence Tomography (OCT) and Optical Coherence Tomography Angiography (OCT-A), as well as measurement of intraocular pressure (IOP) and blood pressure (BP) in sitting and supine positions. No invasive procedures or treatments will be administered. We will be using the standard clinically available software as well as investigational software available for research purposes. The investigational software has been deemed safe by the manufacturer of the device and does not pose any additional risks to patients. Since not every glaucoma patient has high eye pressure (low-tension glaucoma) or has pressure controlled with medication use (so that the untreated eye pressure is now known), glaucoma subjects using intraocular pressure lowering medication and with IOP < 25 mm Hg may be requested to stop their medication for 1 to 3 weeks, by the treating ophthalmologist depending on the class of medication, before being imaged. Risks are small and include IOP elevation. However, glaucoma progression is on the order of months to years, and not days. Subjects will resume using the medication after the research visit is completed.

ELIGIBILITY:
Inclusion:

* Subjects are healthy controls with or without myopia, and patients with or without myopia with a diagnosis of glaucoma, glaucoma suspect and ocular hypertension
* They will be considered if they are above 18 years old.
* There is no upper age limit
* Subject are not restricted by gender, race or ethnicity.

Exclusion:

-Participants with other ocular or systemic conditions and treatment, which may affect visual function, are excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 1995-04; Primary Completion 2030-07 (Estimated); Study Completion 2030-07 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Linda Zangwill, PhD, Principal Investigator — University of California, San Diego
Locations (1):
- UCSD, Hamilton Glaucoma Center, La Jolla, California, United States

REFERENCES:
- [Result] Sample PA, Weinreb RN, Boynton RM. Acquired dyschromatopsia in glaucoma. Surv Ophthalmol. 1986 Jul-Aug;31(1):54-64. doi: 10.1016/0039-6257(86)90051-2. PMID 3529468
- [Result] Weinreb R.N. and Greve E.L. (Eds.). (2004). Glaucoma diagnosis. Structure and function. The Hague, The Netherlands: Kugler Publications.
- [Result] Anderson DR. Standard perimetry. Ophthalmol Clin North Am. 2003 Jun;16(2):205-12, vi. doi: 10.1016/s0896-1549(03)00005-1. PMID 12809158
- [Result] Anderson AJ, Johnson CA. Frequency-doubling technology perimetry. Ophthalmol Clin North Am. 2003 Jun;16(2):213-25. doi: 10.1016/s0896-1549(03)00011-7. PMID 12809159
- [Result] Racette L, Sample PA. Short-wavelength automated perimetry. Ophthalmol Clin North Am. 2003 Jun;16(2):227-36, vi-vii. doi: 10.1016/s0896-1549(03)00010-5. PMID 12809160
- [Result] Zangwill LM, Abunto T, Bowd C, Angeles R, Schanzlin DJ, Weinreb RN. Scanning laser polarimetry retinal nerve fiber layer thickness measurements after LASIK. Ophthalmology. 2005 Feb;112(2):200-7. doi: 10.1016/j.ophtha.2004.08.019. PMID 15691551
- [Result] Medeiros FA, Zangwill LM, Bowd C, Vessani RM, Susanna R Jr, Weinreb RN. Evaluation of retinal nerve fiber layer, optic nerve head, and macular thickness measurements for glaucoma detection using optical coherence tomography. Am J Ophthalmol. 2005 Jan;139(1):44-55. doi: 10.1016/j.ajo.2004.08.069. PMID 15652827
- [Result] Zangwill LM, Chan K, Bowd C, Hao J, Lee TW, Weinreb RN, Sejnowski TJ, Goldbaum MH. Heidelberg retina tomograph measurements of the optic disc and parapapillary retina for detecting glaucoma analyzed by machine learning classifiers. Invest Ophthalmol Vis Sci. 2004 Sep;45(9):3144-51. doi: 10.1167/iovs.04-0202. PMID 15326133
- [Result] Bowd C, Zangwill LM, Medeiros FA, Hao J, Chan K, Lee TW, Sejnowski TJ, Goldbaum MH, Sample PA, Crowston JG, Weinreb RN. Confocal scanning laser ophthalmoscopy classifiers and stereophotograph evaluation for prediction of visual field abnormalities in glaucoma-suspect eyes. Invest Ophthalmol Vis Sci. 2004 Jul;45(7):2255-62. doi: 10.1167/iovs.03-1087. PMID 15223803
- [Result] Sample PA, Chan K, Boden C, Lee TW, Blumenthal EZ, Weinreb RN, Bernd A, Pascual J, Hao J, Sejnowski T, Goldbaum MH. Using unsupervised learning with variational bayesian mixture of factor analysis to identify patterns of glaucomatous visual field defects. Invest Ophthalmol Vis Sci. 2004 Aug;45(8):2596-605. doi: 10.1167/iovs.03-0343. PMID 15277482
- [Result] Medeiros FA, Sample PA, Weinreb RN. Frequency doubling technology perimetry abnormalities as predictors of glaucomatous visual field loss. Am J Ophthalmol. 2004 May;137(5):863-71. doi: 10.1016/j.ajo.2003.12.009. PMID 15126151
- [Result] Medeiros FA, Zangwill LM, Bowd C, Weinreb RN. Comparison of the GDx VCC scanning laser polarimeter, HRT II confocal scanning laser ophthalmoscope, and stratus OCT optical coherence tomograph for the detection of glaucoma. Arch Ophthalmol. 2004 Jun;122(6):827-37. doi: 10.1001/archopht.122.6.827. PMID 15197057
- [Result] Mohammadi K, Bowd C, Weinreb RN, Medeiros FA, Sample PA, Zangwill LM. Retinal nerve fiber layer thickness measurements with scanning laser polarimetry predict glaucomatous visual field loss. Am J Ophthalmol. 2004 Oct;138(4):592-601. doi: 10.1016/j.ajo.2004.05.072. PMID 15488786
- [Result] Belghith A, Medeiros FA, Bowd C, Liebmann JM, Girkin CA, Weinreb RN, Zangwill LM. Structural Change Can Be Detected in Advanced-Glaucoma Eyes. Invest Ophthalmol Vis Sci. 2016 Jul 1;57(9):OCT511-8. doi: 10.1167/iovs.15-18929. PMID 27454660
- [Result] Diniz-Filho A, Abe RY, Zangwill LM, Gracitelli CP, Weinreb RN, Girkin CA, Liebmann JM, Medeiros FA. Association between Intraocular Pressure and Rates of Retinal Nerve Fiber Layer Loss Measured by Optical Coherence Tomography. Ophthalmology. 2016 Oct;123(10):2058-65. doi: 10.1016/j.ophtha.2016.07.006. Epub 2016 Aug 20. PMID 27554036
- [Result] Gracitelli CP, Tatham AJ, Zangwill LM, Weinreb RN, Abe RY, Diniz-Filho A, Paranhos A Jr, Baig S, Medeiros FA. Asymmetric Macular Structural Damage Is Associated With Relative Afferent Pupillary Defects in Patients With Glaucoma. Invest Ophthalmol Vis Sci. 2016 Apr;57(4):1738-46. doi: 10.1167/iovs.15-18079. PMID 27064394
- [Result] Hammel N, Belghith A, Bowd C, Medeiros FA, Sharpsten L, Mendoza N, Tatham AJ, Khachatryan N, Liebmann JM, Girkin CA, Weinreb RN, Zangwill LM. Rate and Pattern of Rim Area Loss in Healthy and Progressing Glaucoma Eyes. Ophthalmology. 2016 Apr;123(4):760-70. doi: 10.1016/j.ophtha.2015.11.018. Epub 2015 Dec 30. PMID 26746597
- [Result] Saunders LJ, Medeiros FA, Weinreb RN, Zangwill LM. What rates of glaucoma progression are clinically significant? Expert Rev Ophthalmol. 2016;11(3):227-234. doi: 10.1080/17469899.2016.1180246. Epub 2016 May 13. PMID 29657575
- [Result] Silverman AL, Hammel N, Khachatryan N, Sharpsten L, Medeiros FA, Girkin CA, Liebmann JM, Weinreb RN, Zangwill LM. Diagnostic Accuracy of the Spectralis and Cirrus Reference Databases in Differentiating between Healthy and Early Glaucoma Eyes. Ophthalmology. 2016 Feb;123(2):408-414. doi: 10.1016/j.ophtha.2015.09.047. Epub 2015 Oct 31. PMID 26526632
- [Result] Skaat A, De Moraes CG, Bowd C, Sample PA, Girkin CA, Medeiros FA, Ritch R, Weinreb RN, Zangwill LM, Liebmann JM; Diagnostic Innovations in Glaucoma Study and African Descent and Glaucoma Evaluation Study Groups. African Descent and Glaucoma Evaluation Study (ADAGES): Racial Differences in Optic Disc Hemorrhage and Beta-Zone Parapapillary Atrophy. Ophthalmology. 2016 Jul;123(7):1476-83. doi: 10.1016/j.ophtha.2016.03.025. Epub 2016 Apr 23. PMID 27117781
- [Result] Suh MH, Zangwill LM, Manalastas PI, Belghith A, Yarmohammadi A, Medeiros FA, Diniz-Filho A, Saunders LJ, Weinreb RN. Deep Retinal Layer Microvasculature Dropout Detected by the Optical Coherence Tomography Angiography in Glaucoma. Ophthalmology. 2016 Dec;123(12):2509-2518. doi: 10.1016/j.ophtha.2016.09.002. Epub 2016 Oct 18. PMID 27769587
- [Result] Suh MH, Zangwill LM, Manalastas PI, Belghith A, Yarmohammadi A, Medeiros FA, Diniz-Filho A, Saunders LJ, Yousefi S, Weinreb RN. Optical Coherence Tomography Angiography Vessel Density in Glaucomatous Eyes with Focal Lamina Cribrosa Defects. Ophthalmology. 2016 Nov;123(11):2309-2317. doi: 10.1016/j.ophtha.2016.07.023. Epub 2016 Aug 31. PMID 27592175
- [Result] Yarmohammadi A, Zangwill LM, Diniz-Filho A, Suh MH, Manalastas PI, Fatehee N, Yousefi S, Belghith A, Saunders LJ, Medeiros FA, Huang D, Weinreb RN. Optical Coherence Tomography Angiography Vessel Density in Healthy, Glaucoma Suspect, and Glaucoma Eyes. Invest Ophthalmol Vis Sci. 2016 Jul 1;57(9):OCT451-9. doi: 10.1167/iovs.15-18944. PMID 27409505
- [Result] Yarmohammadi A, Zangwill LM, Diniz-Filho A, Suh MH, Yousefi S, Saunders LJ, Belghith A, Manalastas PI, Medeiros FA, Weinreb RN. Relationship between Optical Coherence Tomography Angiography Vessel Density and Severity of Visual Field Loss in Glaucoma. Ophthalmology. 2016 Dec;123(12):2498-2508. doi: 10.1016/j.ophtha.2016.08.041. Epub 2016 Oct 7. PMID 27726964
- [Result] Yousefi S, Balasubramanian M, Goldbaum MH, Medeiros FA, Zangwill LM, Weinreb RN, Liebmann JM, Girkin CA, Bowd C. Unsupervised Gaussian Mixture-Model With Expectation Maximization for Detecting Glaucomatous Progression in Standard Automated Perimetry Visual Fields. Transl Vis Sci Technol. 2016 May 3;5(3):2. doi: 10.1167/tvst.5.3.2. eCollection 2016 May. PMID 27152250
- [Result] Zhang C, Tatham AJ, Abe RY, Diniz-Filho A, Zangwill LM, Weinreb RN, Medeiros FA. Corneal Hysteresis and Progressive Retinal Nerve Fiber Layer Loss in Glaucoma. Am J Ophthalmol. 2016 Jun;166:29-36. doi: 10.1016/j.ajo.2016.02.034. Epub 2016 Mar 3. PMID 26949135
- [Result] Zhang C, Tatham AJ, Abe RY, Hammel N, Belghith A, Weinreb RN, Medeiros FA, Liebmann JM, Girkin CA, Zangwill LM. Macular Ganglion Cell Inner Plexiform Layer Thickness in Glaucomatous Eyes with Localized Retinal Nerve Fiber Layer Defects. PLoS One. 2016 Aug 18;11(8):e0160549. doi: 10.1371/journal.pone.0160549. eCollection 2016. PMID 27537107
- [Result] Akagi T, Zangwill LM, Saunders LJ, Yarmohammadi A, Manalastas PIC, Suh MH, Girkin CA, Liebmann JM, Weinreb RN. Rates of Local Retinal Nerve Fiber Layer Thinning before and after Disc Hemorrhage in Glaucoma. Ophthalmology. 2017 Sep;124(9):1403-1411. doi: 10.1016/j.ophtha.2017.03.059. Epub 2017 May 9. PMID 28499748
- [Result] Bowd C, Zangwill LM, Weinreb RN, Medeiros FA, Belghith A. Estimating Optical Coherence Tomography Structural Measurement Floors to Improve Detection of Progression in Advanced Glaucoma. Am J Ophthalmol. 2017 Mar;175:37-44. doi: 10.1016/j.ajo.2016.11.010. Epub 2016 Nov 30. PMID 27914978
- [Result] De Moraes CG, Hood DC, Thenappan A, Girkin CA, Medeiros FA, Weinreb RN, Zangwill LM, Liebmann JM. 24-2 Visual Fields Miss Central Defects Shown on 10-2 Tests in Glaucoma Suspects, Ocular Hypertensives, and Early Glaucoma. Ophthalmology. 2017 Oct;124(10):1449-1456. doi: 10.1016/j.ophtha.2017.04.021. Epub 2017 May 24. PMID 28551166
- [Result] De Moraes CG, Murphy JT, Kaplan CM, Reimann JJ, Skaat A, Blumberg DM, Al-Aswad L, Cioffi GA, Girkin CA, Medeiros FA, Weinreb RN, Zangwill L, Liebmann JM. beta-Zone Parapapillary Atrophy and Rates of Glaucomatous Visual Field Progression: African Descent and Glaucoma Evaluation Study. JAMA Ophthalmol. 2017 Jun 1;135(6):617-623. doi: 10.1001/jamaophthalmol.2017.1082. PMID 28494060
- [Result] Hammel N, Belghith A, Weinreb RN, Medeiros FA, Mendoza N, Zangwill LM. Comparing the Rates of Retinal Nerve Fiber Layer and Ganglion Cell-Inner Plexiform Layer Loss in Healthy Eyes and in Glaucoma Eyes. Am J Ophthalmol. 2017 Jun;178:38-50. doi: 10.1016/j.ajo.2017.03.008. Epub 2017 Mar 16. PMID 28315655
- [Result] Kabbara SW, Zangwill LM, Mundae R, Hammel N, Bowd C, Medeiros FA, Weinreb RN, Belghith A. Comparing optical coherence tomography radial and cube scan patterns for measuring Bruch's membrane opening minimum rim width (BMO-MRW) in glaucoma and healthy eyes: cross-sectional and longitudinal analysis. Br J Ophthalmol. 2018 Mar;102(3):344-351. doi: 10.1136/bjophthalmol-2016-310111. Epub 2017 Aug 3. PMID 28774935
- [Result] Shoji T, Zangwill LM, Akagi T, Saunders LJ, Yarmohammadi A, Manalastas PIC, Penteado RC, Weinreb RN. Progressive Macula Vessel Density Loss in Primary Open-Angle Glaucoma: A Longitudinal Study. Am J Ophthalmol. 2017 Oct;182:107-117. doi: 10.1016/j.ajo.2017.07.011. Epub 2017 Jul 20. PMID 28734815
- [Result] Wu Z, Saunders LJ, Zangwill LM, Daga FB, Crowston JG, Medeiros FA. Impact of Normal Aging and Progression Definitions on the Specificity of Detecting Retinal Nerve Fiber Layer Thinning. Am J Ophthalmol. 2017 Sep;181:106-113. doi: 10.1016/j.ajo.2017.06.017. Epub 2017 Jun 29. PMID 28669780
- [Result] Yarmohammadi A, Zangwill LM, Diniz-Filho A, Saunders LJ, Suh MH, Wu Z, Manalastas PIC, Akagi T, Medeiros FA, Weinreb RN. Peripapillary and Macular Vessel Density in Patients with Glaucoma and Single-Hemifield Visual Field Defect. Ophthalmology. 2017 May;124(5):709-719. doi: 10.1016/j.ophtha.2017.01.004. Epub 2017 Feb 10. PMID 28196732
- [Result] Yarmohammadi A, Zangwill LM, Weinreb RN. Reply. Ophthalmology. 2017 May;124(5):e51. doi: 10.1016/j.ophtha.2016.11.031. No abstract available. PMID 28433140
- [Derived] Mahmoudinezhad G, Moghimi S, Latif K, Brye N, Walker E, Nishida T, Du KH, Gunasegaran G, Wu JH, Liebmann JM, Fazio MA, Girkin CA, Zangwill LM, Weinreb RN. Number of macula optical coherence tomography scans needed to detect glaucoma progression. Br J Ophthalmol. 2025 May 30;109(6):675-681. doi: 10.1136/bjo-2023-324916. PMID 39663002
- [Derived] Mohammadzadeh V, Liang Y, Moghimi S, Xie P, Nishida T, Mahmoudinezhad G, Eslani M, Walker E, Kamalipour A, Micheletti E, Wu JH, Christopher M, Zangwill LM, Javidi T, Weinreb RN. Detection of glaucoma progression on longitudinal series of en-face macular optical coherence tomography angiography images with a deep learning model. Br J Ophthalmol. 2024 Nov 22;108(12):1688-1693. doi: 10.1136/bjo-2023-324528. PMID 39117359
- [Derived] Nishida T, Moghimi S, Gunasegaran G, Walker E, Wu JH, Rahmatnejad K, Zangwill LM, Baxter SL, Weinreb RN. Association between metformin use with circumpapillary retinal nerve fibre layer thickness and capillary vessel density in glaucoma. Br J Ophthalmol. 2024 Dec 17;109(1):45-51. doi: 10.1136/bjo-2023-325035. PMID 38839252
- [Derived] Nishida T, Micheletti E, Latif K, Du KH, Weinreb RN, Moghimi S. Impact of smoking on choroidal microvasculature dropout in glaucoma: a cross-sectional study. BMJ Open Ophthalmol. 2023 Oct;8(1):e001421. doi: 10.1136/bmjophth-2023-001421. PMID 37899137
- [Derived] Mahmoudinezhad G, Nishida T, Weinreb RN, Baxter SL, Chang AC, Nikkhoy N, Walker E, Liebmann JM, Girkin CA, Moghimi S. Associations of smoking and alcohol consumption with the development of open angle glaucoma: a retrospective cohort study. BMJ Open. 2023 Oct 4;13(10):e072163. doi: 10.1136/bmjopen-2023-072163. PMID 37793935
- [Derived] Wu JH, Moghimi S, Nishida T, Walker E, Kamalipour A, Li E, Mahmoudinezhad G, Zangwill LM, Weinreb RN. Evaluation of the long-term variability of macular OCT/OCTA and visual field parameters. Br J Ophthalmol. 2024 Jan 29;108(2):211-216. doi: 10.1136/bjo-2022-322470. PMID 36585126
- [Derived] Mahmoudinezhad G, Moghimi S, Nishida T, Micheletti E, Du KH, Mohammadzadeh V, Wu JH, Kamalipour A, Weinreb RN. Intraocular pressure increases the rate of macular vessel density loss in glaucoma. Br J Ophthalmol. 2024 Jan 29;108(2):181-187. doi: 10.1136/bjo-2022-322261. PMID 36535749
- [Derived] Wu JH, Moghimi S, Nishida T, Mahmoudinezhad G, M Zangwill L, Weinreb RN. Association of macular vessel density and ganglion cell complex thickness with central visual field progression in glaucoma. Br J Ophthalmol. 2023 Nov 22;107(12):1828-1833. doi: 10.1136/bjo-2022-321870. PMID 36150750
- [Derived] Wu JH, Moghimi S, Nishida T, Mohammadzadeh V, Kamalipour A, Zangwill LM, Weinreb RN. Association of macular OCT and OCTA parameters with visual acuity in glaucoma. Br J Ophthalmol. 2023 Nov;107(11):1652-1657. doi: 10.1136/bjo-2022-321460. Epub 2022 Sep 9. PMID 36126109
- [Derived] Nishida T, Moghimi S, Hou H, Proudfoot JA, Chang AC, David RCC, Kamalipour A, El-Nimri N, Rezapour J, Bowd C, Zangwill LM, Weinreb RN. Long-term reproducibility of optical coherence tomography angiography in healthy and stable glaucomatous eyes. Br J Ophthalmol. 2023 May;107(5):657-662. doi: 10.1136/bjophthalmol-2021-320034. Epub 2021 Dec 21. PMID 34933897
- [Derived] Yang Z, Mansouri K, Moghimi S, Weinreb RN. Nocturnal Variability of Intraocular Pressure Monitored With Contact Lens Sensor Is Associated With Visual Field Loss in Glaucoma. J Glaucoma. 2021 Mar 1;30(3):e56-e60. doi: 10.1097/IJG.0000000000001727. PMID 33137021
- [Derived] Hu R, Marin-Franch I, Racette L. Prediction accuracy of a novel dynamic structure-function model for glaucoma progression. Invest Ophthalmol Vis Sci. 2014 Oct 30;55(12):8086-94. doi: 10.1167/iovs.14-14928. PMID 25358735
- [Derived] Balasubramanian M, Arias-Castro E, Medeiros FA, Kriegman DJ, Bowd C, Weinreb RN, Holst M, Sample PA, Zangwill LM. Detecting glaucoma progression from localized rates of retinal changes in parametric and nonparametric statistical framework with type I error control. Invest Ophthalmol Vis Sci. 2014 Mar 19;55(3):1684-95. doi: 10.1167/iovs.13-13246. PMID 24519427
- [Derived] Tatham AJ, Meira-Freitas D, Weinreb RN, Marvasti AH, Zangwill LM, Medeiros FA. Estimation of retinal ganglion cell loss in glaucomatous eyes with a relative afferent pupillary defect. Invest Ophthalmol Vis Sci. 2014 Jan 29;55(1):513-22. doi: 10.1167/iovs.13-12921. PMID 24282221
- [Derived] Lisboa R, Mansouri K, Zangwill LM, Weinreb RN, Medeiros FA. Likelihood ratios for glaucoma diagnosis using spectral-domain optical coherence tomography. Am J Ophthalmol. 2013 Nov;156(5):918-926.e2. doi: 10.1016/j.ajo.2013.06.017. Epub 2013 Aug 20. PMID 23972303
- [Derived] Tatham AJ, Weinreb RN, Zangwill LM, Liebmann JM, Girkin CA, Medeiros FA. Estimated retinal ganglion cell counts in glaucomatous eyes with localized retinal nerve fiber layer defects. Am J Ophthalmol. 2013 Sep;156(3):578-587.e1. doi: 10.1016/j.ajo.2013.04.015. Epub 2013 Jun 7. PMID 23746612
- [Derived] Tatham AJ, Weinreb RN, Zangwill LM, Liebmann JM, Girkin CA, Medeiros FA. The relationship between cup-to-disc ratio and estimated number of retinal ganglion cells. Invest Ophthalmol Vis Sci. 2013 May 7;54(5):3205-14. doi: 10.1167/iovs.12-11467. PMID 23557744
- [Derived] Lisboa R, Paranhos A Jr, Weinreb RN, Zangwill LM, Leite MT, Medeiros FA. Comparison of different spectral domain OCT scanning protocols for diagnosing preperimetric glaucoma. Invest Ophthalmol Vis Sci. 2013 May 13;54(5):3417-25. doi: 10.1167/iovs.13-11676. PMID 23532529
- [Derived] Balasubramanian M, Kriegman DJ, Bowd C, Holst M, Weinreb RN, Sample PA, Zangwill LM. Localized glaucomatous change detection within the proper orthogonal decomposition framework. Invest Ophthalmol Vis Sci. 2012 Jun 14;53(7):3615-28. doi: 10.1167/iovs.11-8847. PMID 22491406
- [Derived] Bowd C, Lee I, Goldbaum MH, Balasubramanian M, Medeiros FA, Zangwill LM, Girkin CA, Liebmann JM, Weinreb RN. Predicting glaucomatous progression in glaucoma suspect eyes using relevance vector machine classifiers for combined structural and functional measurements. Invest Ophthalmol Vis Sci. 2012 Apr 30;53(4):2382-9. doi: 10.1167/iovs.11-7951. PMID 22427577
- [Derived] Medeiros FA, Zangwill LM, Mansouri K, Lisboa R, Tafreshi A, Weinreb RN. Incorporating risk factors to improve the assessment of rates of glaucomatous progression. Invest Ophthalmol Vis Sci. 2012 Apr 24;53(4):2199-207. doi: 10.1167/iovs.11-8639. PMID 22410555
- [Derived] Mansouri K, Leite MT, Weinreb RN, Tafreshi A, Zangwill LM, Medeiros FA. Association between corneal biomechanical properties and glaucoma severity. Am J Ophthalmol. 2012 Mar;153(3):419-427.e1. doi: 10.1016/j.ajo.2011.08.022. Epub 2011 Oct 21. PMID 22018707
- [Derived] Medeiros FA, Leite MT, Zangwill LM, Weinreb RN. Combining structural and functional measurements to improve detection of glaucoma progression using Bayesian hierarchical models. Invest Ophthalmol Vis Sci. 2011 Jul 29;52(8):5794-803. doi: 10.1167/iovs.10-7111. PMID 21693614
- See also: Official website at UCSD — https://shileyeye.ucsd.edu